CLINICAL TRIAL: NCT00146237
Title: Phenytoin as an Augmentation for SSRI Failures: A Controlled Study
Brief Title: Phenytoin as an Augmentation for SSRI Failures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: The Rogosin Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMHC-3581
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Depression
Keywords: phenytoin; SSRI failure; depression
MeSH Terms: conditions — Depression | interventions — Phenytoin

INTERVENTIONS:
Drug: phenytoin

SUMMARY:
About two-thirds of depressed patients respond to a standard course of serotonin specific reuptake inhibitor (SSRI's) within 3-4 weeks. While some clinicians advise continued watchful waiting after this time or switch to a different reuptake-blocker based antidepressant, result of such conservative strategies are usually disappointing. For severe depression electroconvulsive therapy (ECT) is an option and for atypical depressions monoamine oxide inhibitors (MAO) inhibitors often give relief at this point. A unique strategy with both theoretical and practical implications is lithium augmentation (Fava et al, 1994). Addition of lithium to SSRI failures at 3-4 weeks is consistently and sometimes dramatically found to be helpful. This is considered true even by those authors who advocate use of lithium under usual circumstances only in bipolar patients.

Lithium in recent years has been joined as a mood stabilizer by carbamazepine and valproate. Phenytoin, ignored for many years as a possible anticonvulsant mood stabilizer, has been recently reported in double-blind controlled trials to be anti-manic (Mishory et al, 2000) and also prophylactic in BP disorder (Mishory et al, 2003).

Data on mood stabilizers other than lithium as augmentors in SSRI failures are sparse. Carbamazepine (Steinacher et al, 2002) and valproate (Barbee et al, 2002) have been used. Given our recent preliminary results of phenytoin's efficacy in unipolar depression (Nemets et al, 2005) and its analogy to lithium as a mood stabilizer, it seems important to study phenytoin as a possible augmentation of SSRI failures.

We have published a negative study previously of inositol as an augmentation of SSRI failures, enrolling forty-two patients over two years (Nemets et al, 1999). Antidepressant failures are easier to recruit from referring physicians in our center than are untreated patients, whom clinicians are reluctant to refer for new drug studies given the adequacy of standard treatment in 2/3 of them. Thus we estimate that we could enroll 20 patients per year in such a study. Survey of the literature of Li augmentation suggests that 40 phenytoin vs. 40 placebo should give adequate power to detect a significant phenytoin effect if the phenytoin effect is similar to that of lithium.

DETAILED DESCRIPTION:
About two-thirds of depressed patients respond to a standard course of serotonin specific reuptake inhibitor (SSRI's) within 3-4 weeks. While some clinicians advise continued watchful waiting after this time or switch to a different reuptake-blocker based antidepressant, result of such conservative strategies are usually disappointing. For severe depression electroconvulsive therapy (ECT) is an option and for atypical depressions monoamine oxide inhibitors (MAO) inhibitors often give relief at this point. A unique strategy with both theoretical and practical implications is lithium augmentation (Fava et al, 1994). Addition of lithium to SSRI failures at 3-4 weeks is consistently and sometimes dramatically found to be helpful. This is considered true even by those authors who advocate use of lithium under usual circumstances only in bipolar patients.

Lithium in recent years has been joined as a mood stabilizer by carbamazepine and valproate. Phenytoin, ignored for many years as a possible anticonvulsant mood stabilizer, has been recently reported in double-blind controlled trials to be anti-manic (Mishory et al, 2000) and also prophylactic in BP disorder (Mishory et al, 2003).

Data on mood stabilizers other than lithium as augmentors in SSRI failures are sparse. Carbamazepine (Steinacher et al, 2002) and valproate (Barbee et al, 2002) have been used. Given our recent preliminary results of phenytoin's efficacy in unipolar depression (Nemets et al, 2005) and its analogy to lithium as a mood stabilizer, it seems important to study phenytoin as a possible augmentation of SSRI failures.

We have published a negative study previously of inositol as an augmentation of SSRI failures, enrolling forty-two patients over two years (Nemets et al, 1999). Antidepressant failures are easier to recruit from referring physicians in our center than are untreated patients, whom clinicians are reluctant to refer for new drug studies given the adequacy of standard treatment in 2/3 of them. Thus we estimate that we could enroll 20 patients per year in such a study. Survey of the literature of Li augmentation suggests that 40 phenytoin vs. 40 placebo should give adequate power to detect a significant phenytoin effect if the phenytoin effect is similar to that of lithium.

The study has been approved by the Helsinki Committee and all patients must give written informed consent. Patients will be evaluated for study if they meet DSM-IV criteria for major depression without psychotic features. Patients can enter the study if they had at least 3 weeks of treatment with SSRI at clinically adequate doses (150mg fluvoxamine, 20mg fluoxetine, or 20mg paroxetine) and still have a score of at least 18 on the Hamilton Depression Scale (HDS) (on 24 item scale) with at most mild improvement from onset of SSRI treatment. Patients with alcohol or drug abuse or patients with unstable medical illnesses are excluded. Design is parallel double-blind. Patients continue SSRI treatment of the same medication and dose they received before entry. They are randomly assigned to phenytoin or identical placebo capsules. Patients will be rated on the HDRS weekly for four weeks after addition of phenytoin or placebo. Patients who do not improve at least 1 unit on the GCI every two weeks will be dropped from the study for ethical reasons and referred to open treatment. HDRS ratings are done weekly by an experienced psychiatrist (BN) blind to the treatment medication.

Blood levels of phenytoin will be reported by the lab to the treating psychiatrist after "dummy" levels are assigned by the control psychiatrist to patients on placebo.

All patients will be evaluated physically and EKG, liver and kidney functions, and blood cell count performed before entering the study.

Special attention will be given to instruction of patients in dental hygiene and patients showing signs of gingival hyperplasia will be dropped. Studies in epilepsy show that this side effect is surprisingly uncommon, despite wide publicity. No cases were seen in our previous short-term study or prophylactic study (Mishory et al, 2000; Mishory et al, 2003). Nonlinear pharmacokinetics, drug interactions and the consequent danger of toxicity will be handled by careful blood levels monitoring. Patients with significant side effects or toxicity will be dropped from the study. Patients with indications of hypersensitivity reactions (morbilliform rash, Stevens-Johnson syndrome, systemic lupus erythematosus, hepatic necrosis, neutropenia and leukopenia, red-cell aplasia, agranulocytosis, aplastic- or megalo- anemia, or thrombocytopenia) will be dropped from the study.

Importance: Almost one third of patients fail to respond to standard antidepressants. Proof of efficacy of phenytoin augmentation in such cases would: 1) be a useful addition to our clinical armamentarium 2) strengthen the theoretical profile of phenytoin as an antimanic, antidepressant and mood stabilizing compound parallel to lithium and several other anticonvulsants 3) raise useful and heuristic ideas for mechanistic studies of phenytoin's effects on mood.

References

Barbee JG, Jamhour NJ. (2002). Lamotrigine as an augmentation agent in treatment-resistant depression. J Clin Psychiatry 63:737-741.

Fava M, Rosenbaum J, McGrath P, et al. (1994). Lithium and tricyclic augmentation of fluoxetine treatment for resistant major depression. Am J Psychiatry 15:1372-1374.

Mishory A, Yaroslavsky Y, Bersudsky Y, Belmaker RH. (2000). Phenytoin as an antimanic anticonvulsant: a controlled study. American Journal of Psychiatry 157:463-465.

Mishory A, Winokur M, Bersudsky Y.(2003). Prophylactic effect of phenytoin in BP disorder: a controlled study. Bipolar Disorder 5(6):464-7.

Nemets B, Stahal Z, Belmaker RH (2002). Omega-3 fatty acid treatment of depressive breakthrough during unipolar maintenance. American Journal of Psychiatry 159:477-479.

Nemets B, Mishory A, Levine J, Belmaker RH. (1999). Inositol addition does not improve depression in SSRI treatment failures. Journal of Neural Transmission 106:795-798.

Nemets B & Levine J (2005). Phenytoin is equivalent to fluoxetine in unipolar depression: a controlled study 66(5):586-90.

Steinacher L, Vandel P, Zullino DF, CB Eap, Brawand-Amey M, Baumann P. (2002). Carbamazepine augmentation in depressive patients non-responding to citalopram: a pharmacokinetic and clinical pilot study. Eur Neuropsychopharmacol 12:255-260.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-65
* DSM-IV criteria for major depression without psychotic features
* at least 3 weeks of treatment with SSRI at clinically adequate dose with at most mild improvement from onset of SSRI treatment
* Hamilton Depression Scale score of at least 18

Exclusion Criteria:

* ideations of suicide
* pregnancy
* drug or alcohol abuse
* unstable medical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-11; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: RH Belmaker, MD, Study Director — Ben-Gurion University of the Negev
Locations (2):
- Israel (2):
  - Beersheva Mental Health Center, Beersheva
  - Sarah Herzog Memorial Hospital, Jerusalem